CLINICAL TRIAL: NCT00004572
Title: Identification and Therapy Efficacy of Type 2 Diabetes in Hispanic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR02558-0129; M01RR002558 (NIH)
Record Dates: First submitted 2000-02-16; First posted 2000-02-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Defined Population

INTERVENTIONS:
Procedure: Sustacal challenge

SUMMARY:
The two major types of diabetes are type 1 and type 2 diabetes. Although most patients with type 2 diabetes are older than age 40, type 2 diabetes has been reported with increasing frequency among patients under the age of 20. This form of diabetes has been called type 2 diabetes of youth, abbreviated type 2Y. Little is known about the etiology of type 2Y; however, clinicians believe that it occurs most commonly in obese children of particular ethnic groups. A positive family history appears to be one major risk factor for developing type 2Y diabetes. The individual contribution of ethnicity, obesity, and genetics to type 2Y have yet to be elucidated. There is no consensus regarding treatment with type 2Y diabetes. Observation of our Hispanic patients in the Houston area reveals a large number with type 2Y. The major purpose of this study is to examine the genetic and environmental risk factors such as family history, ethnicity, and obesity in Hispanic children with type 2Y diabetes. SPECIFIC AIMS: 1) To examine the genetic and environmental risk factors and clinical signs associated with type 1 diabetes and type 2 diabetes of youth. 2) To compare the efficacy of the treatment modalities, insulin and oral agents, in type 2Y patients. METHODS: We will undertake a retrospective case study, to include a review of hypothesized risk factors in all the medical records of pediatric diabetes patients seen at University of Texas. We anticipate that approximately 200 patients with type 1 diabetes and 30 patients with type 2Y diabetes will be identified. A Sustacal challenge test will be done in patients with a suspected diagnosis of type 2Y in order to confirm the clinical diagnosis. Parents will be contacted by phone for a detailed pedigree intake. Type 1 and type 2Y patients will be compared for each of the studied features. A retrospective review of diabetes type 2 therapies used in type 2Y patients will be undertaken through further examination of the medical records in order to compare insulin treatment to oral agents. We will also test a subset of the patients for the gene identified in adult Hispanics with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Approximately 30 pediatric patients (ages 10-18) believed to have a diagnosis of type 2Y. Each subject must have been diagnosed for at least one year.

Exclusion Criteria:

* Patients over the age of 18 or under the age of 10
* Patients in whom intellectual functioning is impaired sufficiently to interfere with the understanding of the protocol.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult